CLINICAL TRIAL: NCT06158529
Title: A Multicentre Clinical Study of High-frequency Electrical Spinal Cord Stimulation Versus Electrical Spinal Cord Stimulation in the Treatment of Diabetic Peripheral Neuropathic Pain
Brief Title: High-frequency SCS Versus SCS in the Treatment of Diabetic Peripheral Neuropathic Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fan BiFa (Other)
Collaborators: Peking University Third Hospital (Other); Xuanwu Hospital, Beijing (Other); Civil Aviation General Hospital (Other); Shenzhen Sixth People's Hospital (Other); Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor-Investigator, Fan BiFa, China-Japan Friendship Hospital, China-Japan Friendship Hospital
Organization: China-Japan Friendship Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SF-2022-1-4061
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Painful Diabetic Peripheral Neuropathy
Keywords: spinal cord stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- spinal cord stimulation (Active Comparator): Traditional spinal cord electrical stimulation
  Interventions: Device: spinal cord stimulator
- high frequency spinal cord stimulation (Experimental): High frequency SCS (HF-SCS) technology can treat chronic pain without relying on the tingling sensation
  Interventions: Device: high frequency spinal cord stimulation

INTERVENTIONS:
Device: spinal cord stimulator — A spinal cord stimulator is an implanted device that sends low levels of electricity directly into the spinal cord to relieve pain.
  Arms: spinal cord stimulation
Device: high frequency spinal cord stimulation — A spinal cord stimulator is an implanted device that sends low levels and high frequency of electricity directly into the spinal cord to relieve pain.
  Arms: high frequency spinal cord stimulation

SUMMARY:
Application of High-Frequency Spinal Cord Stimulation (HF-SCS) in the Treatment of Painful Diabetic Peripheral Neuropathy (PDPN): A multicenter, randomized controlled study comparing its clinical efficacy with traditional spinal cord stimulation for PDPN. The study aims to observe the impact of HF-SCS on the neurological function and microcirculation of PDPN patients, elucidating the correlation between the underlying diabetes and the efficacy of HF-SCS therapy on PDPN. The goal is to enhance the treatment standards for PDPN, improve the quality of life for this population, and overall treatment outcomes. Simultaneously, the study aims to contribute evidence-based medicine for the mechanistic exploration of PDPN.

DETAILED DESCRIPTION:
The incidence rate of diabetes peripheral neuropathic pain (DPNP) is high, and there is no clear and effective treatment, which is a clinical problem to be solved urgently.

Traditional spinal cord electrical stimulation (SCS) has the potential to treat DPNP, and its efficacy depends on the tingling sensation generated by the electrical stimulation covering the painful area of the patient. The neurological dysfunction of DPNP patients and the defects of traditional SCS lead to unsatisfactory therapeutic effects.

The emerging high-frequency SCS (HF-SCS) technology can treat chronic pain without relying on tingling sensation. Multiple evidence shows that HF-SCS has better long-term efficacy in treating chronic neuropathic pain than traditional SCS.

Our research group has also preliminarily confirmed the effectiveness and safety of HF-SCS in treating DPNP.

Therefore, this study intends to use a multicenter prospective randomized controlled clinical research method to explore the superiority of HF-SCS in treating DPNP compared to traditional SCS, and establish a standardized diagnosis and treatment platform database for DPNP in Beijing.

This project will provide high-level evidence-based medicine for the treatment of DPNP with HF-SCS, and also provide clinical big data support for the standardized diagnosis and treatment of DPNP in the future.

On the basis of medical engineering integration, an innovative remote control system is applied to achieve real-time adjustment and precise regulation of SCS treatment parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with diabetes, aged between 18 and 80 years old;
2. Symmetrical pain in the distal lower extremities with or without dysesthesia;
3. Duration of symptoms exceeding 6 months;
4. Pain described as stabbing and/or electric shock-like and/or burning sensation;
5. Abnormal Quantitative Sensory Testing (QST);
6. Presence of hyperalgesia and allodynia;
7. Absence of lower limb reflexes and muscle strength abnormalities;
8. Normal MRI or CT scans without spinal canal stenosis or other spinal abnormalities.

Exclusion Criteria:

1. Concurrent severe cardiovascular and cerebrovascular diseases;
2. History of lumbar spine surgery, trauma, or spinal canal stenosis within the past 6 months, or a history of lumbar spine surgery, trauma, or spinal canal stenosis that would impact the SCS surgery and pain assessment in this study;
3. Presence of radicular symptoms;
4. Other spinal abnormalities, such as benign or malignant tumors, congenital abnormalities of the spine, spinal instability, etc.;
5. Coexisting disorders of the coagulation system, malignant tumors, infections, and psychiatric or psychological disorders;
6. Pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
treatment effectiveness | 3months
  The treatment effectiveness is assessed based on the reduction of Numeric Rating Scale (NRS) scores for pain three months after treatment compared to before treatment. Specifically, a decrease of ≥50% in the pain NRS score [(NRS score at 3 months post-treatment - NRS score before treatment) / NRS score before treatment] ≥ 50% is considered the criterion for treatment effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: BiFa Fan, master, Study Chair — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No